CLINICAL TRIAL: NCT01141751
Title: A Phase IV, Observational, Open-label, Multi-center Comparison Study of the Newly Developed and Validated MusiQoL (Multiple Sclerosis International Quality of Life Questionnaire) Instrument With the Health-related QoL (MSQOL-54) Questionnaire in Subjects With Relapsing Forms of Multiple Sclerosis (RMS*) on Rebif® Therapy
Brief Title: An Observational Study Comparing Multiple Sclerosis International Quality of Life Questionnaire (MusiQoL) and Multiple Sclerosis Quality of Life-54 Instrument (MSQOL-54) in Relapsing Multiple Sclerosis (RMS) Patients on Long-term Rebif® Therapy
Acronym: COMPARE
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: 00066
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2013-06

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple sclerosis; Expanded Disability Status Scale; Multiple Sclerosis, Relapsing-Remitting; Rebif; Beta-1, interferon
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Significant data from placebo-controlled clinical trials have demonstrated the efficacy of Rebif in relapsing remitting multiple sclerosis (RRMS) with reduction in relapse rate, delay in disability progression, and reduction in magnetic resonance imaging (MRI) activity and accumulation of lesion burden. Multiple sclerosis (MS), a chronic neurological diseases, can have diverse effects on the lives of subjects and their families. In controlled clinical trials, clinical measurement in MS has focused on impairments of neurological assessment using Expanded Disability Status Score (EDSS). The assessment of the impact of MS on the non-physical aspect of dysfunction is not often measured, or reported. Furthermore, traditional clinical measures have not been able to assess the effects of neurological illness on quality of life (QoL), which is becoming an increasingly important topic to neurologists treating subjects with varied neurological conditions.

This observational, one arm, multicentric study is aimed to assess the usefulness of the Multiple Sclerosis International Quality of Life Questionnaire (MusiQoL) instrument in comparison with the Multiple Sclerosis Quality of Life-54 instrument (MSQOL-54 questionnaire) in RMS subjects on Rebif therapy and to assess the effectiveness of Rebif therapy using health related quality of life (HRQoL) measures.

DETAILED DESCRIPTION:
Multiple sclerosis is a chronic, inflammatory, demyelinating disease of the central nervous system (CNS) and is one of the most common causes of neurological disability in young adults. The neuropathology of the disease is marked by accumulation of leukocytes in the CNS, oligodendrocyte loss, demyelination, axonal atrophy, and neuronal loss. Clinically it is characterized by multi-focal recurrent attacks of neurological symptoms and signs with variable recovery and eventually, the majority of subjects develop a progressive clinical course of MS. The exact cause of MS is unknown, although an autoimmune process has been implicated. Genetic susceptibility plays a role in disease initiation but unidentified environmental factors may also be involved. Three clinical forms of MS are recognized: primary progressive multiple sclerosis (PPMS), secondary progressive multiple sclerosis (SPMS) and RRMS. Primary progressive subjects are characterized by slow and steady accumulation of neurological deficits from onset without superimposed attacks. Subjects with RRMS have exacerbations or relapses with subsequent variable recovery (remission). Secondary progressive multiple sclerosis is characterized by the steady accumulation of significant and persistent neurological deficit with or without superimposed relapses.

The concept of quality of life (QoL) is defined by the World Health Organization (WHO) as an individual's perception of his or her life within the cultural context and value system in which he or she lives, in respect to objectives, expectations, norms and worries. It is a very complex and broad concept, influenced at various levels by the subject's physical health state, psychological health state, level of independence, social relations and relationship with the overall surrounding environment. A critical element of HRQoL is that it reflects the subject's assessment of the impact of his/her illness, not the physician's perspective. Professional interest in the concept of QoL has increased over the course of the past years, particularly within the framework of health care programs for chronic diseases. Health related quality of life measures can be subdivided into generic and disease-specific measures. Generic measures are designed to assess subjects with diverse medical conditions and they may not capture all relevant aspects of a specific illness. However, disease-specific measures developed from generic HRQoL tools may not truly reflect perspectives from the subjects with specific diseases. The MusiQoL questionnaire is a subject focused questionnaire being developed by an independent scientific steering committee in conjunction with MS subjects, neurologists, and health economists since 2000.

OBJECTIVES

* To assess the usefulness of MusiQoL in clinical practice in comparison with the established disease specific QoL instrument MSQOL-54
* To evaluate the effectiveness of Rebif therapy with respect to HRQoL in a longitudinal study in subjects with RMS

This is an observational, one arm, multicentric study. Quality of life data from the MusiQoL instrument and MSQOL-54 questionnaire, as well as physical health outcomes such EDSS, will be collected bi-annually in subjects with RMS.

ELIGIBILITY:
Inclusion Criteria:

* Subjects eligible for Rebif therapy according to indications and clinical use in the Rebif Product Monograph (and subject who agreed to start on Rebif therapy)
* Subjects who have read, understood, signed and dated the informed consent form

Exclusion Criteria:

* Subjects who are unable to fill in the questionnaires by him/herself
* Subjects who have used disease modifying drugs within the last month (or 30 days) prior to study Day 1

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with RMS who are eligible for Rebif therapy in Canada
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2005-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Usefulness of MusiQoL in clinical practice in comparison with the established disease specific QoL instrument MSQOL-54 | Baseline to 24 months (or Early Termination)
  The usefulness of the MusiQoL versus the MSQOL-54 questionnaire will be evaluated based on the numbers of missing items; the difficulty of completing each instrument; responses to a subject evaluation questionnaire (the proportion of subjects who prefer MusiQoL versus MSQOL-54 according to their assessment of the best user-friendly QoL questionnaire, time spent to complete each questionnaire and references of the subjects according to the evaluation questionnaire); subject's QoL instrument rating assessed with a VAS (visual analogue scale, ranged from 0 to 10)

SECONDARY OUTCOMES:
Evaluation of QoL instrument scores between baseline and month 24 and the relationship to measures of disease activity (relapses) and disease severity (EDSS) | Baseline to 24 months (or Early Termination)
Relationship between Folstein mini-mental status examination (MMSE) and Frontal assessment battery (FAB) scores and QoL instrument scores | Baseline to 24 months (or Early Termination)
Relationship between depression score and QoL instrument scores | Baseline to 24 months (or Early Termination)
Number of relapses | Baseline to 24 months (or Early Termination)
Expanded Disability Status Score (EDSS) scores | Baseline to 24 months (or Early Termination)
Number of progressions on the EDSS score | Baseline to 24 months (or Early Termination)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono, a division of EMD Inc., Canada

REFERENCES:
- [Derived] Vickrey BG, Lee L, Moore F, Moriarty P. EDSS Change Relates to Physical HRQoL While Relapse Occurrence Relates to Overall HRQoL in Patients with Multiple Sclerosis Receiving Subcutaneous Interferon beta -1a. Mult Scler Int. 2015;2015:631989. doi: 10.1155/2015/631989. Epub 2015 Jul 5. PMID 26236506